CLINICAL TRIAL: NCT07016529
Title: Diagnostic Utility of Myeloperoxidase for Differentiating Irritable Bowel Syndrome From Inflammatory Bowel Disease in Patients With Lower GIT Symptoms
Brief Title: Diagnostic Study for Differentiating Functional From Organic Diseases in Patients With Lower GIT Symptoms
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rania Mohammad Abd-ellatif, Internal medicine resident, Sohag University
Other Study IDs: Soh-Med--25-5-9MS
Record Dates: First submitted 2025-05-28; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome (IBS); Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group "normal": normal individuals
- case group 1 "patients with lower GIT symptoms suggestive of irritable bowel syndrome": those who fulfill the criteria of irritable bowel disease.no intervention needed.
- case group 2 "patients with lower GIT symptoms suggestive of inflammatory bowel disease": those with bloody diarrhea or chronic diarrhea or other manifestations suggest inflammatory bowel disease.no intervention needed.

SUMMARY:
The study is intended to find a new trusted, cost-effective biomarker for differentiating irritable bowel syndrome from inflammatory bowel disease to decrease the use of unnecessary invasive methods in patients with irritable bowel syndrome

DETAILED DESCRIPTION:
Myeloperoxidase is a lysosomal protein that is released from granules of neutrophil granulocytes during inflammation. the study design relies on the fact that there is no mucosal inflammation in case of functional gastrointestinal tract (GIT) disorders like irritable bowel syndrome (IBS), but organic gastrointestinal conditions like inflammatory bowel diseases (IBD) has mucosal inflammation and neutrophil influx into the mucosa.

the study is designed to assess myeloperoxidase levels in both conditions and assessing its reliability in differentiation between them.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) presenting with chronic lower gastrointestinal symptoms, such as diarrhea, abdominal pain, or altered bowel habits, for a duration exceeding 6 weeks.
* Patients with no prior diagnosis of IBD or IBS.
* Patients willing to provide informed consent and comply with study requirements.
* Those without recent use of immunosuppressants or anti-inflammatory medications that could affect biomarker levels

Exclusion Criteria:

* Patients with a confirmed diagnosis of IBD and currently on treatment.
* Those with acute gastroenteritis, infectious colitis, or positive stool cultures for pathogens.
* Patients diagnosed with colorectal cancer, celiac disease, or other known organic GI disorders.
* Recent antibiotic, NSAID, or corticosteroid use within the past 4 weeks.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with lower GIT symptoms seeking medical advice at Department of Internal Medicine, Gastroenterology Outpatient Clinic, Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
efficacy of myeloperoxidase for differentiating irritable bowel syndrome from inflammatory bowel disease. | baseline
  Number of patients with elevated myeloperoxidase in irritable bowel syndrome and those with inflammatory bowel disease.

IPD SHARING:
Plan to Share IPD: Undecided